CLINICAL TRIAL: NCT05204875
Title: Functional Lung Imaging in Patients With Respiratory Compromise Undergoing Endobronchial Valve Placement
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Temple University (Other)
Collaborators: Respiratory Compromise Institute (Unknown)
Responsible Party: Sponsor
Other Study IDs: 269649
Record Dates: First submitted 2021-12-22; First posted 2022-01-24 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Emphysema
MeSH Terms: conditions — Emphysema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Functional lung imaging: Assess the applicability of XV ventilation distribution and heterogeneity for BLVR candidate screening compared to conventional tools of quantitative HRCT and ventilation perfusion scanning.
  Interventions: Radiation: X-ray Velocimetry

INTERVENTIONS:
Radiation: X-ray Velocimetry — X-ray Velocimetry (XV) technology images the motion of the lungs, determines airway volumes and measures regional lung ventilation during spontaneous breathing.

SUMMARY:
Bronchoscopic lung volume reduction (BLVR) using endobronchial valves is effective in improving quality of life in patients suffering from emphysema. BLVR treatment in advanced emphysema requires targeted segmental or sub-segmental placement of endobronchial valves (EBV) to achieve total lobar occlusion to induce effective lobar volume reduction. BLVR procedure success rate declines in patients with incomplete lobar fissure integrity due to the potential for collateral ventilation to circumvent EBV lobar occlusion. Current methods that assess lobar collateral ventilation as a correlate of fissure integrity are imperfect, resulting in a significant percentage of patients having equivocal assessment, leading to suboptimal selection of patients and potential for inappropriate selection of patients for BLVR. Additionally, methods used to select the target lobe for EBV placement predominately rely on the extent of emphysematous destruction. There is also a need to select based on the extent of physiological disturbance at the lobar level. Distribution of ventilation or regional ventilation heterogeneity may be associated with collateral ventilation. Therefore, in this study we wish to quantify lobar distribution of ventilation and ventilation heterogeneity in patients undergoing investigation for BLVR to determine the additive contribution of functional lung imaging for assessing lobar physiological derangement and suitability for EBV treatment.

DETAILED DESCRIPTION:
Approach: A novel functional lung imaging, X-ray Velocimetry (XV) technology images the motion of the lungs, determines airway volumes and measures regional lung ventilation during spontaneous breathing. Specific measurements of lobar volume at end inspiration, expiration and the tidal breathing changes, inspiratory and expiratory lobar flow and estimation of airway flow resistance using x-ray velocimetry. These variables will be used to explore indices related to collateral ventilation by comparing time-volume changes based on segmentation and differential residual. The performance of XV has been assessed in cohort and case series of patients undergoing therapy for cancer, demonstrating changes in ventilation distribution and heterogeneity. The objective of the current investigation is to determine whether XV technology can assist in determining lobar selection, indicators of success, or response-related clinical outcomes with BLVR.

Scope: Examine ventilation distribution and heterogeneity using XV functional lung imaging analysis in moderate to severe COPD undergoing evaluation for BLVR.

Aims: 1) Assess the applicability of XV ventilation distribution and heterogeneity for BLVR candidate screening compared to conventional tools of quantitative HRCT and ventilation perfusion scanning.

2) Identify characteristics of lobar ventilation distribution and ventilation heterogeneity in candidates being assessed for BLVR.

3) Determine whether if there is an association between functional lung imaging data and clinical status (6MWD, St George's Questionnaire, CAT, mMRC (Modified Medical Research Council) Dyspnea Scale).

Study Design:

a. Participant Recruitment This is an adaptive trial design in 10 patients in consecutive recruitment at Temple University Hospital. As subsequent sites initiate investigation, a small number of roll-in study participants (n=2) will be enrolled for site validation. Patient managed by Temple University Hospital with inclusion criteria will be identified by Dr. Gerard Criner for possible inclusion in this study. A waiver for informed consent will be obtained to allow review of their medical records to determine if these patients may be eligible for study inclusion. It is anticipated that most of these patients will have known underlying lung disease. The patient will be screened by the principal investigator or designee for eligibility. Upon meeting all eligibility criteria, the patient will be approached by the principal investigator or designee to obtain informed consent for inclusion into the study. Discussion of the study will take place in a private room and will include the relevance of this study, risks they may encounter, data collected, and the protection of their personal information.

All those included in the study will have a diagnosis consistent with existing or potential clinical work up for BLVR procedure. As this is a cross-sectional study subjects will not be randomized. The study timeframe for participation will be defined as the time beginning from recruitment for participation in functional lung imaging which is adjunct measurement to an existing clinical procedure, until the collection of all data associated with the study. Data may be collected from medical records whilst the study is approved by the IRB. The clinical course will neither depend upon, be altered by nor rely on any of the research data collected as part of this study. To examine the relationship of study data with standard of care, clinical status, disease exacerbation, prior history of hospitalization, the data collection period will include historical health records and lung health records before and after the functional lung imaging scan

ELIGIBILITY:
Inclusion Criteria:

* Emphysema
* Undergoing evaluation and planned treatment with BLVR
* Adults, 40 years of age and older
* Consents to functional lung imaging evaluation
* Access to previous chest CT as part of the clinical workup for BLVR

Exclusion Criteria:

* Known contraindication to BLVR
* Currently receiving mechanical ventilation, intensive or other critical care
* Pregnant women
* Contraindication to ionizing radiation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COPD undergoing bronchoscopic lung volume reduction
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-07-05 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The objective of the current investigation is to determine whether XV technology can assist in determining lobar selection, indicators of success, or response-related clinical outcomes with BLVR. | functional lung imaging and software analysis will be available after the procedure
  Functional lung imaging analysis in endobronchial valve placement

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Criner, MD, Principal Investigator — Temple University
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States